CLINICAL TRIAL: NCT03867721
Title: The Preference of Neuromuscular Patients Regarding Available Equipment for Daytime Mouthpiece Ventilation: a Randomized Cross-over Study
Brief Title: Patient Preference for Mouthpiece Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Revalidatieziekenhuis InkendaaI (Network)
Responsible Party: Principal Investigator, Kristien Mostinckx, Head of Rehabilitation Department, Revalidatieziekenhuis InkendaaI
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: 2014-WMT-001
Record Dates: First submitted 2019-03-03; First posted 2019-03-08 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Neuromuscular Diseases
Keywords: noninvasive ventilation
MeSH Terms: conditions — Neuromuscular Diseases | interventions — Ventilators, Mechanical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ventilator PB560 (Covidien) (Experimental): The non-dedicated (NON-DED) set comprised a ventilator for MPV (PB560) using a single active tubing with an exhalation valve. A custom-made arm support and plastic mouthpiece were used.
  Interventions: Device: Ventilator
- Ventilator Trilogy (Philips Respironics) (Experimental): The dedicated (DED) set comprised a ventilator for MPV (Trilogy 100, Philips Respironics; with dedicated software, with a single passive tubing without exhalation valve. A back-up rate set at zero cycle per minute was associated with a kiss trigger, with a smart flexible tube support system and with a silicone made mouthpiece designed as a straw.
  Interventions: Device: Ventilator

INTERVENTIONS:
Device: Ventilator — Comparison of two ventilators for mouthpiece ventilation

SUMMARY:
BACKGROUND:

Patients with severe neuromuscular disorders (NMDs) are likely to develop progressive respiratory insufficiency, leading to noninvasive ventilation during the night and, later, during night and day. Ventilation via a mouthpiece (MPV) is an elegant option to offer daytime ventilation. The patient preference regarding the ideal material for daytime MPV is unclear.

OBJECTIVES:

The purpose of this study was to determine which ventilator, tubing support and mouthpiece was most effective and preferred by patients with NMDs.

METHODS:

Two separate MPV equipment sets were compared in 20 patients with NMDs in a randomized cross-over study. The first set consisted in a non-dedicated ventilator for MPV (PB560, Covidien) combined with a customized tubing support on the shoulders and a plastic angled mouthpiece. The second set included an MPV-dedicated ventilator (Trilogy 100, Philips Respironics) without back-up rate and kiss trigger combined with a commercially available tubing support and a silicone straw mouthpiece. The Borg dyspnea score, the free time without noninvasive ventilation, the transcutaneous oxygen saturation (SpO2) and carbon dioxide tension (TcCO2) were recorded without and with MPV. A 17-items list assessing the patient perception about MPV sets was completed.

DETAILED DESCRIPTION:
Materials and Methods

Aims

The primary aim of the study was to compare blood gas measurements, dyspnea score and general perception between the two sets for MPV. The second aim of the study was to determine the preference of patients on MPV equipment according to their free time. We also aimed at collecting individual comments of patients regarding their experience with the two ventilators, arm supports and mouthpieces.

Patients

All individuals affected by NMDs attending our Centre for Home Mechanical Ventilation between 2015 and 2018 who required daytime MPV as an extension of nocturnal NIV were considered for study inclusion. Our criterion for implementing daytime ventilation was the combined presence of increasing dyspnea and increasing workload on inspiratory muscles during the daytime (C) or, ultimately, daytime hypercapnia in the evening when patients lay in bed before starting nocturnal NIV and sleeping (M). All patients used Volume-Assisted Pressure Control mode (VAPC) at night via a Covidien Puritan Bennett PB560 ventilator (Covidien, Mansfield, USA).

Exclusion criteria comprised patients with ineffective NIV during sleep as assessed by the measurement of TcCO2>49mmHg (S), patients with uncontrollable oral leaks with MPV or episode of acute respiratory infection during the trials. The current study was approved by the local ethics committee and registered (N° registered study. Clinical trial.org follows). The patients gave their written informed consent before study inclusion.

Study design

The study design consisted in a randomized cross-over study. Patients served as their own control. Measurements were made during a 48-hour hospitalization that is scheduled every 6 months in patients attending our Centre for Home Mechanical Ventilation. Hospitalization systematically included nocturnal recordings of transcutaneous carbon dioxide tension (TcCO2) and pulse oximetry (SpO2). Randomized trials were decided by toss and tested during a 1-hour session of assisted breathing via MPV on two separate days. Patients were seated in their wheelchair and trials started with connecting patients to transcutaneous TcCO2 and SpO2 measurements.

Equipment for MPV

Two different MPV equipment sets were compared (figure 1). Each set included separate ventilators, tubing supports and mouthpieces. Both ventilators used volume assisted control mode (VAC) according to the patient preference reported in a previous study (Q).

The first set consisted in a non-dedicated (NON-DED) ventilator for MPV (PB560) using a single active tubing with an exhalation valve. The trigger was set on high sensitivity. Solutions to avoid nuisance from disconnection alarms were used according to a report from Boitano and colleagues (O). The PB560 was combined with a local custom-made tubing support in thermo-formable plastic U-piece placed on the patient shoulders (figure 1 A) described in a previous report (M). The mouthpiece consisted in a 22mm white angled hard plastic mouthpiece (Philips Respironics; Murrysville, USA). Despite being a non MPV-dedicated set, the NON-DED set was previously reported as safe and an effective (M).

The second set included an MPV-dedicated (DED) ventilator (Trilogy 100, Philips Respironics; Murrysville, USA) with an MPV dedicated software with disconnection alarms switched off. This set included a single passive tubing without exhalation valve. A back-up rate set at zero cycle per minute was associated with a kiss trigger. The kiss trigger consisted in a sensitive flow detection system allowing on-demand ventilation via a constant airflow produced by the ventilator. When this constant flow was disrupted by the engagement and disengagement of the patient's lips from the mouthpiece, a single inspiratory cycle was triggered. Finally, the DED equipment included a smart flexible tube support system attached via a wedge on the patient's wheelchair (figure 1 B). The tubing ended with a silicone made mouthpiece designed as a straw. The backup rate in de DED equipment was copied from nighttime values. Similar VAC mode, tidal volumes and inspiratory times were used in both equipment's to facilitate further comparison. Trials were a succession of intermittent disconnections-reconnections to the mouthpiece. All patients were encouraged to manage leaks around the mouthpiece according to their breathing comfort.

Measurements

Day 1

Forced vital capacity (FVC), maximal inspiratory (MIP) and expiratory pressures (MEP) were measured on the first day in seated position as per ATS/ERS guidelines (T) via a heated Fleisch no. 2 pneumotachometer (Metabo, Lausanne, Switzerland). The Borg dyspnea scale on 10 points reflecting the degree of comfortable breathing was also recorded on the first day (C). Other daytime baseline measurements such as transcutaneous oxygen saturation (SpO2) and carbon dioxide tension (TcCO2) were recorded without daytime ventilation via an ear clip connected to a Sentec monitoring (SenTec AG, Therwil, Swizerland). This technique was validated for continuous monitoring of PaCO2 during sleep in this group of patients (U). The participants were asked to determine their free time defined as the time of comfortable spontaneous breathing without NIV. Finally, the maximal active mouth opening (space between upper and lower teeth) was measured.

Day 2 and 3

The maximal TcCO2 and minimal SpO2 values obtained during the trials were measured. As in day 1, the Borg dyspnea score was recorded to evaluate the breathing comfort during MPV trials. A 17-items list assessing the patient perception with a Likert scale ranging from 0 to 5 (0: maximal dissatisfaction, 5: maximal satisfaction) was completed during the trials.

ELIGIBILITY:
Inclusion Criteria:

* All individuals affected by NMDs attending our Centre for Home Mechanical Ventilation between January 2015 and December 2018 who required daytime MPV as an extension of nocturnal NIV

Exclusion Criteria:

* Patients with no need for daytime ventilation
* patients with ineffective NIV during sleep as assessed by the measurement of TcCO2>49mmHg (S)
* patients with uncontrollable oral leaks with MPV or episode of acute respiratory infection during the trials

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Transcutaneous Carbon dioxyde | Day 2: continuous recording during trial 1 (30min)
  Maximal level of CO2 tension in blood (PCO2)
Transcutaneous Carbon dioxyde | Day 3: continuous recording during trial 2 (30min)
  Maximal level of CO2 tension in blood (PCO2)
Trancutaneous Oxygen saturation | Day 2: continuous recording during trial 1 (30min)
  Minimal level of Oxygen saturation (SpO2)
Trancutaneous Oxygen saturation | Day 3: continuous recording during trial 2 (30min)
  Minimal level of Oxygen saturation (SpO2)
Borg dyspnea score | Day 2: at the end of trial 1
  Score (0-10 points; 0: very comfortable; 10: very uncomfortable) to evaluate the subjective feeling of breathing comfort. Borg is not an abbreviation but it is name of the author who validated the score. Dyspnea score is named "Borg" visual analogic score
Borg dyspnea score | Day 3: at the end of trial 2
  Score (0-10 points; 0: very comfortable; 10: very uncomfortable) to evaluate the subjective feeling of breathing comfort. Borg is not an abbreviation but it is name of the author who validated the score. Dyspnea score is named "Borg" visual analogic score
A 17-item questionnaire assessing the patient perception | Day 2: at the end of trial 1
  Score (0-5 points; 0: very bad ; 10: very good ) to evaluate the subjective perception (easiness-comfort) of patients with the ventilator equipment.
A 17-item questionnaire assessing the patient perception | Day 3: at the end of trial 2
  Score (0-5 points; 0: very bad ; 10: very good ) to evaluate the subjective perception (easiness-comfort) of patients with the ventilator equipment.

SECONDARY OUTCOMES:
Freetime | On day 1 (baseline)
  Time of comfortable spontaneous breathing without assisted ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- Michel Toussaint, Vlezenbeek, Belgium

IPD SHARING:
Plan to Share IPD: No